CLINICAL TRIAL: NCT05357443
Title: Effect of Vagus Nerve Preservation During Gastric Bypass on Gastrin Level and Marginal Ulcer Formation
Brief Title: SH Dr. Chen Gastric Bypass Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanford Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SH Gastric Bypass Study
Record Dates: First submitted 2022-04-19; First posted 2022-05-02 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Gastric Bypass
MeSH Terms: interventions — Gastric Bypass

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric Bypass with Transection of Vagal Nerves (Active Comparator)
  Interventions: Procedure: Gastric bypass with transection of vagal nerves
- Gastric Bypass Without Transection of Vagal Nerves (Placebo Comparator)
  Interventions: Procedure: Gastric bypass without transection of vagal nerves

INTERVENTIONS:
Procedure: Gastric bypass with transection of vagal nerves — Vagal nerve interruption above the level of the stomach is a known treatment for complicated peptic ulcer disease. It is not commonly performed during routine gastric bypass. The vagi are, however, interrupted part-way down the stomach to create the gastric pouch. This is the pars flaccida technique.
  Arms: Gastric Bypass with Transection of Vagal Nerves
Procedure: Gastric bypass without transection of vagal nerves — Dissection between the neurovascular bundle and the stomach, spareing the vagus nerves. This is the perigastric technique.
  Arms: Gastric Bypass Without Transection of Vagal Nerves

SUMMARY:
Evaluation of serum gastrin levels and their effect on marginal ulcer formation.

DETAILED DESCRIPTION:
Prospective, randomized, interventional trial. Participants will be randomized to one of two surgical techniques, either with transection of the vagal nerves, or without. Outcomes including compare marginal ulcer rates will be compared using serum gastrin levels before and after surgery and gastric pH during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of obesity or disorder of metabolism undergoing routine gastric bypass surgical intervention
* Capable of giving signed informed consent.

Exclusion Criteria:

* Under 18 years of age
* Ineligible for gastric bypass surgery
* Pregnant women or women actively seeking to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Marginal Ulcer | From surgical intervention to five years after surgery
  Number of participants with a change in serum gastrin levels compared pre- and post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sugong Chen, MD, Principal Investigator — Sanford Health
Locations (1):
- Sanford Health, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No